CLINICAL TRIAL: NCT05766839
Title: A 2-Part, Open-Label, Phase 2, Multiple Dose Study to Evaluate the Pharmacodynamic Effects, Safety, and Tolerability of Patiromer in Children Under 12 Years of Age With Hyperkalaemia (EMERALD2)
Brief Title: Patiromer for Treatment of Hyperkalaemia in Children Under 12 Years of Age
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vifor Pharma, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLY5016-208p; 2023-505252-21-00 (Other: EU CT Number)
Record Dates: First submitted 2023-01-19; First posted 2023-03-13 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — patiromer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patiromer (Experimental): 4-week pharmacodynamic /dose-ranging period
  Cohort 1: 6 to less than (<)12 years of age
  Cohort 2: 2 to <6 years of age
  Cohort 3: 0 to <2 years of age; In Cohort 3, a minimum of 3 study participants will be assessed in the subgroup of 0 to <6 months and another 3 study participants in the subgroup 6 to <24 months of age.
  Interventions: Drug: Patiromer

INTERVENTIONS:
Drug: Patiromer — Patiromer will be given once daily; In Cohort 3, depending on the dose and the study participant's age, the total daily dose might be split

SUMMARY:
A study to evaluate the pharmacodynamic effects, safety, and tolerability of patiromer in children under 12 years of age with hyperkalaemia.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria must be met for each participant:

* Paediatric participants (<12 years of age) with hyperkalaemia at screening.
* Participant's age should not reach 12 years during the 28 days of the pharmacodynamic/dose-ranging period.
* Participant is able to receive regular external feeding and medication, including via tubes, i.e., percutaneous endoscopic gastrostomy (PEG) or entero-gastric feeding tube.
* At screening/baseline, the results from 2 separate and consecutive potassium assessments using the same measurement method (whole blood, plasma, or serum) need to be above the age-appropriate upper limit of normal (ULN).
* If taking any renin-angiotensin aldosterone system inhibitors (RAASi), beta blockers, fludrocortisone, or diuretic medications, must be on a stable dose for at least 14 days prior to screening.
* Parent(s) or legally authorised representative(s) or another appropriate person delegated by the legally authorised representatives must be available to help the study-site personnel ensure follow-up; accompany the participant to the study site on each assessment day; accurately and reliably dispense investigational product as directed.
* Females of childbearing potential must be non-lactating, must have a negative pregnancy test at screening, and must have used an effective, acceptable form of contraception (e.g., abstinence) for at least 1 month before patiromer administration. Females of childbearing potential must agree to continue using contraception throughout the study and for 1 month after the last dose of patiromer.
* If undergoing peritoneal dialysis, participants must be on a stable treatment plan for a minimum of 4 weeks prior to screening, or at least 8 weeks prior to screening if newly initiated on peritoneal dialysis.

Exclusion Criteria:

The following criteria exclude a participant from participating in this trial:

* Preterm birth infants with <37 weeks of gestation cannot be included in Cohort 3.
* Participants who due to their general condition, e.g., anaemia or low body weight, are not suitable to have blood volume withdrawn.
* Any of the following renal conditions: maintenance haemodialysis, renal artery stenosis, and acute kidney injury (defined by 2012 Kidney Disease Improving Global Outcomes) or a history of acute renal insufficiency in the past 3 months. Note: Chronic kidney disease (CKD) is not excluded.
* A history of or current diagnosis of a severe gastrointestinal (GI) diagnosis or surgery that could affect GI transit of the drug (delayed gastric emptying), such as a severe swallowing disorder, severe gastroesophageal reflux, uncorrected pyloric stenosis, intussusception, any other intestinal obstruction (e.g., Hirschsprung disease, chronic intestinal pseudo-obstruction, clinically significant postsurgical abdominal adhesions) or any gut-shortening surgical procedure prior to screening. Pre-gastric above-mentioned pathologies may be disregarded in case of existence of a PEG or entero-gastric feeding tube, as the PEG or entero-gastric feeding tube will serve for nutrition and investigational product administration.
* Active cancer, currently on cancer treatment, or history of cancer in the past 2 years (except for non-melanoma skin cancer).
* Scheduled for kidney transplant procedure during the first 28 days after Day 1.
* History of sudden infant death in a sibling (only for participants <2 years of age at screening).
* Use of the following medications if doses have not been stable for at least 14 days prior to screening or if doses are anticipated to change during the 4-week pharmacodynamic/ dose-ranging period: digoxin, bronchodilators, theophylline, heparins (including low molecular heparins), tacrolimus, mycophenolate mofetil, cyclosporine, trimethoprim, or cotrimoxazole.
* Use of any investigational product for an unapproved indication within 30 days prior to screening or within 5 half-lives, whichever is longer.
* Known hypersensitivity to patiromer or its components.
* If the child is being breastfed:

  1. There is suspicion of current alcohol or substance misuse/abuse in breastfeeding mother
  2. The breastfeeding mother is taking potassium supplements

Other protocol defined Inclusion/Exclusion criteria may apply

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in potassium levels (mmol/L) | From baseline to Day 28
  May be measured as serum, plasma, whole blood, potassium

SECONDARY OUTCOMES:
Change in potassium levels (mmol/L) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
  May be measured as serum, plasma, whole blood, potassium
Occurrence of treatment-emergent adverse events (TEAEs) | Part 1: Day 1 up to end of treatment (Day 28 ±3 Days); Part 2: Day 1 up to follow-up visit (Up to 54 weeks)
Occurrence of serious adverse events (SAEs) | Part 1: Day 1 up to end of treatment (Day 28 ±3 Days); Part 2: Day 1 up to follow-up visit (Up to 54 weeks)
Change from baseline in resting heart rate (beats per minute) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in systolic blood pressure (mmHg) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in diastolic blood pressure (mmHg) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in body temperature (Celsius) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Number of patients with ECG abnormalities | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in chemistry laboratory evaluation: Calcium (mg/dL) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in chemistry laboratory evaluation: Phosphate (mg/dL) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in chemistry laboratory evaluation: Magnesium (mg/dL) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in chemistry laboratory evaluation: Potassium (mEq/L) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in chemistry laboratory evaluation: Sodium (mEq/L) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in chemistry laboratory evaluation: Creatinine (mg/dL) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in chemistry laboratory evaluation: Serum bicarbonate (mEq/L) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in chemistry laboratory evaluation: Blood urea nitrogen (mEq/L) | From baseline to Day 3, Day 7, Day 14, Day 28, and during Part 2: up to 52 weeks
Change from baseline in haematology laboratory evaluation: White blood cells (10^9/L) | From baseline to Day 7, Day 14, Day 28, and EoT visit for Part 2 (week 52)
Change from baseline in haematology laboratory evaluation: Red blood cells count (10^12/L) | From baseline to Day 7, Day 14, Day 28, and EoT visit for Part 2 (week 52)
Change from baseline in haematology laboratory evaluation: Haemoglobin (10^12/L) | From baseline to Day 7, Day 14, Day 28, and EoT visit for Part 2 (week 52)
Change from baseline in haematology laboratory evaluation: Haematocrit (%) | From baseline to Day 7, Day 14, Day 28, and EoT visit for Part 2 (week 52)
Change from baseline in haematology laboratory evaluation: Platelet count (10^9/L) | From baseline to Day 7, Day 14, Day 28, and EoT visit for Part 2 (week 52)
Change from baseline in haematology laboratory evaluation: Blood fluoride (ng/mL) | From baseline to Day 7, Day 14, Day 28, and EoT visit for Part 2 (week 52)
Occurrence of blood potassium below the lower limit of normal (LLN) (mmol/L) | Part 1: Screening up to end of treatment (Day 28 ±3 Days); Part 2: Day 1 up to end of treatment (Up to 52 weeks)
Occurrence of blood potassium above the upper limit of normal (ULN) (mmol/L) | Part 1: Screening up to end of treatment (Day 28 ±3 Days); Part 2: Day 1 up to end of treatment (Up to 52 weeks)
Occurrence of blood magnesium at levels specified in protocol (mmol/L) | Part 1: Screening up to end of treatment (Day 28 ±3 Days); Part 2: Day 1 up to end of treatment (Up to 52 weeks)
Occurrence of abnormal clinical laboratory value findings | Part 1: Screening up to end of treatment (Day 28 ±3 Days); Part 2: Day 1 up to end of treatment (Up to 52 weeks)
  Occurrence of clinical laboratory value findings that are outside of normal range of the respective age for: serum calcium, phosphate, fluoride, creatinine, bicarbonate, and blood urea nitrogen levels

CONTACTS AND LOCATIONS:
Overall Officials: Julian Platon, MD, PhD, Study Director — Vifor Pharma, Inc.
Locations (36):
- United States (13):
  - Children's Hospital Colorado Site 84014, Aurora, Colorado
  - UF Health Pediatric Multispecialty Center Site 84006, Jacksonville, Florida
  - Miller School of Medicine, University of Miami Site 84003, Miami, Florida
  - Arnold Palmer Hospital for Children Site 84010, Orlando, Florida
  - Augusta University - Children's Hospital of Georgia Site 84015, Augusta, Georgia
  - University of Illinois College of Medicine Site 84012, Peoria, Illinois
  - Boston Children's Hospital Site 84008, Boston, Massachusetts
  - Children's Mercy Hospitals and Clinics Site 84004, Kansas City, Missouri
  - Duke University Hospital & Medical Center Site 84002, Durham, North Carolina
  - Duke University Hospital Site 84002, Durham, North Carolina
  - The Children's Hospital of Philadelphia Site 84007, Philadelphia, Pennsylvania
  - Vanderbilt Children's Hospital Neurology Site 84013, Nashville, Tennessee
  - Texas Tech University Health Sciences Center Amarillo Site 84009, Amarillo, Texas
- Australia (2):
  - The Royal Children's Hospital (RCH) Site 03601, Parkville
  - Children's Hospital Westmead Centre for Kidney Research Site 03602, Westmead
- Belgium (2):
  - Universitair Ziekenhuis Gent Site 05601, Ghent
  - UZ Leuven Site 05602, Leuven
- Helsingin Yliopistollinen Keskussairaala Uusi Lastensairaala Site 24601, Helsinki, Finland
- France (3):
  - CHRU Montpellier - Arnaud de Villeneuve Site 25001, Montpellier
  - Assistance Publique-Hopitaux de Paris Robert-Debre Site 25003, Paris
  - Hôpital des Enfants - Toulouse Site 25002, Toulouse
- Greece (2):
  - Ippokratio Thessaloniki General Hospital Site 30002, Thessaloniki, Thessaloniki
  - Pan and Aglaia Kyriakou Children's Hospital Site 30001, Athens
- Israel (2):
  - Shaare Zedek Medical Center Site 37602, Jerusalem
  - Schneider Children's Medical Center of Israel Site 37601, Petach Tikvah
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Site 38002, Milan
  - IRCCS Ospedale Pediatrico Bambino Gesù Site 38001, Rome
- Helse Bergen HF Haukeland Universitetssjukehus Site 57801, Bergen, Norway
- Uniwersytecki Szpital Kliniczny we Wrocławiu Site 61601, Wroclaw, Poland
- Unidade Local de Saude de Santo Antonio, E.P.E. Site 62001, Porto, Portugal
- Sidra Medicine Site 63401, Doha, Qatar
- Spitalul Clinic de Urgenta pentru Copii Louis Turcanu Timisoara Site 64201, Timișoara, Romania
- Saudi Arabia (3):
  - King Saud University Site 68202, Riyadh
  - King Faisal Specialist Hospital & Research Centre Site 68201, Riyadh
  - King Abdulaziz Medical City Site 68203, Riyadh
- Al Jalila Children's Hospital Site 78401, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
CSL Vifor acknowledges the importance of data transparency and commits to sharing, upon request from qualified scientific researchers, patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials for medicines and indications approved in the United States (US) and the European Union (EU).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data from Vifor Pharma sponsored non-interventional and interventional clinical trials (phase 1-4) for medicines and indications approved in the US and the EU, will be shared if the evaluation of the request is positive and two years have elapsed since study completion or termination of the program.
Access Criteria: Data is shared upon request from qualified scientific researchers under the prerequisite that the trial subjects' rights are kept fully protected, in particular with regards to Good Clinical Practice and Data Privacy, that the proposed analyses aim to yield an appropriate and valid scientific output and are not in conflict with the publication plan for the study. Requests should be submitted including a description of the data requested, a rationale for the proposed research, a Statistical Analysis Plan, a Publication Plan, qualifications and experience of the research team, disclosure of any conflicts of interests and competitive use of data, and source of research funding. If after evaluation the request is approved, the process of sharing the requested data will be initiated. As a prerequisite, a signed personal data processing and transfer agreement between Vifor Pharma and the data requestor is required.